CLINICAL TRIAL: NCT05655039
Title: The Effect of Pre-rehabilitation and Rehabilitation Period on Functional Status in Inpatient Stroke Patients
Status: Completed | Type: Observational
Sponsor: Sisli Hamidiye Etfal Training and Research Hospital (Other)
Responsible Party: Principal Investigator, Aylin Ayyıldız, Director, Sisli Hamidiye Etfal Training and Research Hospital
Other Study IDs: 2022
Record Dates: First submitted 2022-11-20; First posted 2022-12-16 (Actual); Last update posted 2022-12-16 (Actual); Status verified 2022-12

CONDITIONS: Stroke; Rehabilitation
MeSH Terms: conditions — Stroke | interventions — Rehabilitation

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Rehabilitation — Stroke Rehabilitation Program

SUMMARY:
Patients who underwent inpatient rehabilitation for the last 5 years were retrospectively scanned. The pre-rehabilitation and rehabilitation periods of the patients were determined. At the beginning and end of rehabilitation, patients were evaluated with the Brunsstrom, Barthel and Stroke Impact Scale. The effect of the specified durations on these scales was investigated.

ELIGIBILITY:
Inclusion Criteria:

* 40-90 years old
* Have hemodynamic stability to participate in rehabilitation
* Having had an ischemic or hemorrhagic stroke

Exclusion Criteria:

* Having a serious comorbidity that may preclude rehabilitation
* Malignancy
* Aphasia
* Having a serious perception problem or psychiatric illness
* Having a history of stroke

Ages: 40 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: 40-90-year-old post-stroke patients
Sampling Method: Non-Probability Sample
Enrollment: 108 (Actual)
Dates: Start 2022-09-15 (Actual); Primary Completion 2022-10-15 (Actual); Study Completion 2022-10-15 (Actual)

PRIMARY OUTCOMES:
Brunnsstrom Stages | immediately after Rehabilitation
  The Brunnstrom stages of stroke recovery, or Brunnstrom approach, outlines how spasticity and involuntary motor patterns improve. Minimum score is 1, maximum score is 6. Higher score means better outcome.
Barthel Index | immediately after Rehabilitation
  The Barthel scale is an ordinal scale used to measure performance in activities of daily living. Each performance item is rated on this scale with a given number of points assigned to each level or ranking. It uses ten variables describing ADL and mobility. Minimum score is 0, maximum score is 100. Higher score means better outcome.
Stroke Impact Scale | immediately after Rehabilitation
  The Stroke Impact Scale (SIS) is a self-report questionnaire that evaluates disability and health-related quality of life after stroke. Minimum score is 0, maximum score is 100. Higher score means better outcome.

CONTACTS AND LOCATIONS:
Overall Officials: Banu Kuran, Professor, Study Director — Şişli Hamidiye Etfal Training and Research Hospital
Locations (1):
- University of Health Sciences, Şişli Hamidiye Etfal Training and Research Hospital, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided